CLINICAL TRIAL: NCT04997694
Title: The Effect Of Pre-Surgery Actıve And Passıve Heatıng On Post-Operatıve Hypothermıa, Lıfe Fındıngs And Temperature Comfort
Brief Title: Effect of Preoperative Active Warming and Passive Warming Methods on Perioperative Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Refiye Akpolat, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000-0001-8907-0651
Record Dates: First submitted 2021-06-23; First posted 2021-08-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Hypothermia; Perioperative Care; Vital Signs; Rewarming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: 3 Group randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Heating Group (Experimental): When the participants comes to the preoperative unit before the operation, vital signs, temperature comfort perception scale and shivering level, temperature and humidity measurements of the room are measured by the investigator and Personal Information Form Vital Signs Follow-up Form, Temperature Comfort Perception Scale- The form was recorded in the Shivering Level Diagnosis Form Filling.Before anesthesia was given, heating was performed with the 3M Bair Hugger Model 775 Heating Unit, which has an active heating system, for 20 minutes. The participants, whose surgery was completed, was taken to the postoperative recovery unit, where the vital signs, tremor level, temperature and humidity of the room were measured by the investigator and the Personal Information Form Vital Signs Follow-up Form Shivering Level Diagnosis Form was recorded. One participant was followed every 15 minutes until the body temperature reached 36 0C.
  Interventions: Procedure: Pre Heating
- Pasive Heating Group (Experimental): When the participants comes to the preoperative unit before the operation, vital signs, temperature comfort perception scale and shivering level, temperature and humidity measurements of the room are measured by the investigator and Personal Information Form ,Vital Signs Follow-up Form, Temperature Comfort Perception Scale. The form was recorded in the Shivering Level Diagnosis Form . Before anesthesia was given, heating was performed with a wool blanket, which is a passive heating method, for 20 minutes. The participants, whose surgery was completed, was taken to the postoperative recovery unit, where the vital signs, tremor level, temperature and humidity of the room were measured by the investigator and the Personal Information Form Vital Signs Follow-up Form , Shivering Level Diagnosis Form was recorded. One participant was followed every 15 minutes until the body temperature reached 36 0C.
  Interventions: Procedure: Pre Heating
- Control Group (No Intervention): When the participants comes to the preoperative unit before the operation, vital signs, temperature comfort perception scale and shivering level, temperature and humidity measurements of the room are measured by the investigator and Personal Information Form Vital Signs Follow-up Form , Temperature Comfort Perception Scale The form was recorded in the Shivering Level Diagnosis Form the participants, whose surgery was completed, was taken to the postoperative recovery unit, where the vital signs, tremor level, temperature and humidity of the room were measured by the investigator and the Personal Information Form , Vital Signs Follow-up Form , Shivering Level Diagnosis Form was recorded. One participant was followed every 15 minutes until the body temperature reached 36 0C.

INTERVENTIONS:
Procedure: Pre Heating — Before anesthesia was given, the participants were warmed for 20 minutes with prewarming techniques. Presence of postoperative hypothermia, vital signs and temperature comfort level were evaluated.
  Other Names: Pre Warming
  Arms: Active Heating Group; Pasive Heating Group

SUMMARY:
70% of surgical interventions are abdominal surgeries. Open abdominal surgery is performed in patients for whom minimally invasive approaches are not suitable. In these surgeries in which general anesthesia is used, the duration of the operation is longer, complications are more frequent, and postoperative recovery occurs later. Low body temperature before surgery, preoperative fasting and fluid deprivation before anesthesia, exposure of large body surface areas, evaporative heat loss during skin preparation using volatile solutions, large open cavity or abdominal surgery longer operative time and exposure to anesthesia, during surgical intervention excessive blood loss etc. surgical intervention poses a risk for the formation of undesirable hypothermia.

Cardiovascular and respiratory system problems that may increase mortality due to hypothermia in surgical patients; may cause a decrease in heart rhythm, cardiac output, blood pressure and oxygen saturation, and an increased risk of cardiac arrest and ischemia. With the development of shivering, oxygen consumption increases and the "thermal comfort" of the patient deteriorates. The length of stay in the postoperative unit and hospital stay are prolonged, causing an increase in costs.

Among the rapid recovery protocols, it is recommended to pre-warm the patients in the preoperative period to maintain normothermia. Many complications are prevented by different methods and warming procedures performed in the perioperative period.

In our study, it was aimed to compare the effects of active and passive warming on hypothermia, vital signs and warmth comfort in the postoperative period in patients who will undergo open abdominal surgery.

DETAILED DESCRIPTION:
Before starting the research, permission was obtained from Çukurova University Medical Faculty Balcalı Hospital General Surgery Department Academic Committee and Operating Room Committee, from Balcalı Hospital Chief Physician (Annex-11), and Çukurova Ethics Committee by the investigator . University Faculty of Medicine Non-Interventional Research Ethics Committee approval was received with the date and number of 10.04.2020/98-29 An application was made to the Scientific Research Projects Unit to support the project with all permissions. It has been approved as a Scientific Research Project.

In accordance with the results of the power analysis using the G power 3.1.9.2 program, it was planned to include 30 participants in the active warming group, 30 partici in the passive warming group and 30 participants in the control group, and a simple randomization method was used in the distribution. Sample for study groups Research data were collected in the operating room preoperative unit and postoperative unit between July 2020 and December 2020.

When the participants came to the preoperative unit before the operation, his vital signs, temperature comfort perception scale and shivering level, temperature and humidity of the room were measured by the investigator and recorded in the Personal Information Form, Vital Signs Monitoring Form, Temperature Comfort Perception Scale Form, Shivering Level Diagnostic Form. Before anesthesia was given, one group was heated with the 3M Bair Hugger Model 775 Heating Unit (Hot Air Blowing Warmer Blanket) with an active heating system and the other group with a passive heating system (wool blanket) for 20 minutes, routine application was made to the control group participants by the investigator . Vital signs, tremor levels and temperature comfort perception measurements were made at the 0th, 15th, and 30th minutes in the postoperative unit of the participants after the operation by the investigator . Statistical analyzes of the collected data were made using a package program called SPSS (IBM SPSS Statistics 24). Frequency tables and descriptive statistics were used to interpret the findings. In accordance with parametric methods, the "ANOVA" test (F-table value) was used to compare the measurement values of three or more independent groups, and the "RepeatedMeasures" test (F-Table) was used to compare the measurement values of three or more dependent groups. The "Mann-Whitney U" test (Z-table value) and the "Kruskal-Wallis H" test (χ2- table value) were used to compare the measurement values of two independent groups in accordance with non-parametric methods. ) method was used. "Wilcoxon" test (Z-table value) to compare measurement values of two dependent groups, "Friedman" test (χ2-table value) to compare measurement values of three or more dependent groups, "Pearson-χ2 To examine the relationships between two qualitative variables used "cross tables" were used.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older,
2. Patients with ASA III and below,
3. Under elective general anesthesia, will undergo Open Abdominal Surgery,
4. BMI of 18.5- 29.9 kg/m2,
5. Without neurological, psychiatric, neuromuscular disease,
6. Not addicted to alcohol and drugs,
7. Not mentally retarded,
8. Does not use drugs that will affect thermoregulation such as vasodilators,
9. No history of thyroid disease,
10. Absence of body temperature of 36 0C and 37.5 0C on the morning of the operation,
11. No complication developed during the surgical intervention and no blood transfusion was performed.

Exclusion Criteria:

1. Refusal to participate in the research
2. Complication developed during the operation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
changes in body temperature preheating process | 30 minutes
  The sample size was calculated by performing G-power power analysis. Pre-application measurements and 0., 15., 30. after application. Considering the temperature changes observed in the measurements obtained per minute, the effect size was found to be 0.1844. Accordingly, the number of samples required to achieve 90% power at α=0.05 level was calculated as 78 patients, including at least 26 active warming groups, 26 passive warming groups, and 26 control groups. In order to increase the power of the research, the study was conducted with a total of 90 patients, 30 from each group.
  Participants with a body temperature below 36 0C were considered to be in hypothermia. Non-contact thermometer was used to measure body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Refiye Akpolat, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Sariçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akpolat R, Arslan S. Effect of Prewarming on Postoperative Hypothermia, Vital Signs, and Thermal Comfort: A Randomized Controlled Trial. Ther Hypothermia Temp Manag. 2024 Jun;14(2):89-98. doi: 10.1089/ther.2023.0017. Epub 2023 Jun 16. PMID 37327382